CLINICAL TRIAL: NCT01154543
Title: A Single Center, Open Label, Longitudinal Single Arm Study to Compare the Efficacy and Safety of Prophylactic Famciclovir 500 mg b.d. in HIV Positive Adults With Recurrent Genital Herpes.
Brief Title: Safety and Efficacy of Famciclovir in HIV1 Positive Adults With Recurrent Genital Herpes
Status: Completed | Type: Observational
Sponsor: Holdsworth House Medical Practice (Other)
Responsible Party: Principal Investigator, Dr. Mark Bloch, Dr Mark Bloch, Holdsworth House Medical Practice
Other Study IDs: Famvir™ 500 in HIV
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: HIV Positive; Herpes Simplex, Genital
Keywords: Recurrent genital Herpes Simplex Virus
MeSH Terms: conditions — HIV Seropositivity; Herpes Genitalis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- HIV positive, gential HSV,Famvir™ 500mg bd, suppressive

SUMMARY:
To determine the efficacy of Famvir 500mg bd as suppressive antiviral therapy for acute genital Herpes simplex virus (HSV) outbreaks in HIV subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide signed informed consent
* Documented HIV infection
* In general good health, without other serious medical conditions as deemed by the investigator
* Male or female over 18 years of age
* Diagnosed genital HSV (clinical or laboratory)
* Life expectancy of 12 months or longer per investigator's judgment
* Stable on Famvir 500 mg bd for at least 30 days at time of screening

Exclusion Criteria:

* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>5)mIU/mL).
* Women of childbearing potential who are unwilling to use reliable contraception for the duration of the study.
* History of hypersensitivity to Famvir, its constituents or penciclovir
* Current use of another antiherpetic medication
* Recent history of alcohol or drug abuse, which in the opinion of the investigator may interfere with their compliance with study requirements, or who have any other conditions which in the opinion of the investigator would interfere with the successful completion of study procedures
* Disorder or condition that could interfere with drug absorption, distribution, metabolism or excretion
* Known or suspected to have or past history of renal dysfunction requiring a dosage modification of Famvir 500 bd

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 50-60 patients attending Holdsworth House Medical Practice in Darlinghurst, Sydney, New South Wales with documented HIV-1 infection who are taking Famciclovir 500mg bd as suppressive therapy for management of genital HSV infection who agree to participate in this study will be enrolled after signing HREC approved informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2008-03; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To determine the incidence of acute genital HSV outbreaks whilst taking Famciclovir 500 mg bd during the study period (24 months) | 24 months
  To determine the incidence of acute genital HSV outbreaks whilst taking Famciclovir 500 mg bd during the study period (24 months)and to determine the safety of Famciclovir 500mg bd in this population

SECONDARY OUTCOMES:
To determine the acceptability of Famciclovir 500 mg bd as long term suppressive antiviral therapy | 24 months
  To determine the acceptability of Famciclovir 500 mg bd as long term suppressive antiviral therapy To determine virological & immunological parameters of HIV whilst taking Famciclovir 500 mg as suppressive antiviral therapy To determine patient adherence to Famciclovir 500 mg bd over the study period To determine the incidence of oral HSV outbreaks in subjects taking Famciclovir 500 mg bd as suppressive antiviral therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Bloch, MBBS, Principal Investigator — Australian Health Practitioners Regulation authority